CLINICAL TRIAL: NCT06481735
Title: A Phase 1/2 Multicenter Study Evaluating the Safety and Efficacy of TCR Reserved and Power3 (SPPL3) Gene Knock-out Allogeneic CD19-targeting CAR-T Cell Therapy in Adults With Refractory/Relapsed B-cell Acute Lymphoblastic Leukaemia
Brief Title: TCR Reserved and Power3 (SPPL3) Gene Knock-out Allogeneic CD19-targeting CAR-T Cell Therapy in r/r B-ALL
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Chinese PLA General Hospital (Other)
Collaborators: Peking University (Other)
Responsible Party: Principal Investigator, Han weidong, Director of Biotherapeutic Department, Chinese PLA General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHN-PLAGH-BT-087
Record Dates: First submitted 2024-06-22; First posted 2024-07-01 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Acute Lymphocytic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — fludarabine; fludarabine phosphate; Injections; Cyclophosphamide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with refractory or relapsed B-ALL (Experimental): A conditioning chemotherapy regimen of fludarabine and cyclophosphamide will be administered followed by investigational treatment, Power3 (SPPL3) Gene Knock-out Allogeneic CD19-targeting CAR-T.
  Interventions: Biological: TCR reserved and Power3 (SPPL3) Gene Knock-out Allogeneic CD19-targeting CAR-T cell; Drug: Fludarabine; Drug: Cyclophosphamide

INTERVENTIONS:
Biological: TCR reserved and Power3 (SPPL3) Gene Knock-out Allogeneic CD19-targeting CAR-T cell — Phase 1 dose escalation (3+3) : dose 1 (1 × 10^6 cells/kg) , dose 2 (3 × 10^6 cells/kg), dose 3 (6 × 10^6 cells/kg); Phase 2 : dose of RP2D.
  Other Names: Allogeneic Power3 (SPPL3) knock-out CD19 CAR-T
Drug: Fludarabine — Intravenous fludarabine 30~50 mg/m^2/day on days -5, -4, and -3.
  Other Names: Fludarabine Phosphate for Injection
Drug: Cyclophosphamide — Intravenous cyclophosphamide 500~1000 mg/m^2/day on days -5, -4, and -3.
  Other Names: Cyclophosphamide for Injection

SUMMARY:
The safety and efficacy of the chimeric antigen receptor (CAR)-T, a CD19-targeting, TRAC and Power3 (SPPL3) double gene deleted allogeneic CAR-T cell product, are undergoing rigorous evaluation in non-Hodgkin's lymphoma (NHL) subjects from the ATHENA trial (NCT06014073). Unexpectedly, expansion of the initial residual CD3-positive CAR T from products were measured in patients' peripheral blood (PB) without exception. Accompanying with host immune reconstitution and appearance of the detectable B cells, the CD3-positive allogenic CAR T cells exhibited a compelling amplification advantage over CD3-negative CAR T cells. The amplification of CD3-positive CAR T cell population dynamically suppressed host B cell recovery, and presumably surveilled the recurrence or progression of tumors, but did not induce typical Graft-versus-host-disease (GvHD). Additionally, a series of in vitro experiments illustrated that the HLA-mismatched fratricide between host T cells and TCR-reserved Power3 (SPPL3)-deleted allogenic CAR T cells was markedly slashed, which in combination with investigators' observed clinical safety data supported the notion that only genomic deletion of Power3 (SPPL3) gene in allo-CAR T cells is sufficient to overcome GvHD and host T cell-mediated rejection response.

In this study, investigators will disable the Power3 (SPPL3) gene of T cells from healthy donors to prepare CAR T cells. This approach harnesses the tonic signaling of CAR T cells, resulting in enhanced persistence and improved response to treatment. The purpose of this study is to evaluate the safety and efficacy of allogeneic Power3 (SPPL3) knock-out CD19 CAR-T in B-cell acute lymphoblastic leukaemia (B-ALL).

DETAILED DESCRIPTION:
Phase 1 (dose escalation)

In phase 1, 6-18 subjects will be enrolled. Subjects will receive 3 doses of allogeneic Power3 (SPPL3) knock-out CD19 CAR-T cell therapy ( 1 × 10^6 cells/kg、3 × 10^6 cells/kg、6 × 10^6 cells/kg) increases from low dose to high dose according to the "3 + 3" principle:

Three (3) subjects are enrolled in a cohort corresponding to a dose level. If 1 subject in a cohort of 3 subjects experiences a dose-limiting toxicity (DLT), 3 additional subjects will be enrolled at the current dose level. For safety purposes, the administration of allogeneic Power3 (SPPL3) knock-out CD19 CAR-T will be staggered by 28 days between the first two subjects in each cohort. And for each of the remaining cohorts, the administration of allogeneic Power3 (SPPL3) knock-out CD19 CAR-T will be staggered by 28 days before enter into the next cohort.

Phase 2 (expansion cohort)

In phase 2, 10 to 12 subjects will be enrolled and receive cell infusion at dose of recommended phase 2 dose (RP2D), which will be determined based on the maximum tolerated dose (MTD), occurrence of DLT, the obtained efficacy results, pharmacokinetics/pharmacodynamics and other data according to the phase 1.

Objectives

The primary objectives of the phase 1 were to evaluate the tolerability and safety of allogeneic Power3 (SPPL3) knock-out CD19 CAR-T in patients with refractory/relapsed (r/r) B-ALL, and determine RP2D. The primary purpose of the phase 2 study was to evaluate the efficacy of allogeneic Power3 (SPPL3) knock-out CD19 CAR-T in the above population.

ELIGIBILITY:
Inclusion Criteria:

1. Age 16-70 (inclusive).
2. Patient with r/r CD19+ B-ALL, as per guidelines (NCCN, 2019)

   * For patients with bone marrow involvement, morphologically confirmed with ≥ 5% leukaemic blasts in the bonemarrow.
   * Definition of relapsed disease: Bone marrow or extramedullary relapse after achieving CR with initial treatment, or any bone marrow or extramedullary relapse after allogeneic hematopoietic stem cell transplantation (allo-HSCT).
   * Refractory disease is defined by not achieving an initial CR after 2 cycles of a standard chemotherapy regimen (primary refractory). Subjects who were refractory to subsequent chemotherapy regimens after an initial remission were considered chemorefractory.
3. Toxicities due to prior therapy must be stable and recovered to ≤ Grade 1 (except for hematological toxicities and clinically non-significant toxicities such as alopecia).
4. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2.
5. Adequate renal, hepatic, pulmonary and cardiac function defined as:

   * Serum creatinine≤1.5 upper limit of normal (ULN) or creatinine clearance (as estimated by Cockcroft Gault) ≥ 60 mL/min.
   * Serum alanine aminotransferase / aspartate aminotransferase (ALT/AST) ≤ 3 upper limit of normal (ULN); Total bilirubin ≤ 1.5 ULN, except in subjects with 3) Gilbert's syndrome.
   * Cardiac ejection fraction ≥ 50%, no evidence of pericardial effusion as determined by an echocardiogram (ECHO), and no clinically significant electrocardiogram (ECG) findings.
   * Coagulation Function: International Normalized Ratio (INR) ≤ 1.5 times the upper limit of normal (ULN), and Activated Partial Thromboplastin Time (APTT) ≤ 1.5 times ULN.
   * Baseline oxygen saturation >91% on room air.
6. Subjects of both genders who are willing to practice birth control from the time of consent through 6 months after the completion of conditioning chemotherapy. Females of childbearing potential must have a negative serum or urine pregnancy test (females who have undergone surgical sterilization or who have been postmenopausal for at least 2 years are not considered to be of childbearing potential).
7. Voluntarily participate in this clinical trial and sign an informed consent form.

Exclusion Criteria:

1. Expected survival time < 3 months per Principal Investigator's opinion.
2. History of malignancy other than nonmelanoma skin cancer or carcinoma in situ (e.g. cervix, bladder, breast) unless disease free for at least 3 years.
3. Patients who received any immunocellular or HSCT therapy within 3 months before enrollment.
4. Active central nervous system (CNS) leukaemia (CNS-3).
5. Clinically active significant CNS dysfunction.
6. Known history of irreversible severe neurological toxicity related to previous antileukaemic treatment leading to organic central nervous system lesions.
7. Use of previous anti-leukemic therapy within 5 half-lives prior to allogeneic Power3 (SPPL3) knock-out CD19 CAR-T administration; participation in non-interventional registries or epidemiological studies is allowed.
8. Radioimmunotherapy, radiotherapy, within 8 weeks (except prophylaxis of CNS involvement) before Inclusion.
9. History of severe immediate hypersensitivity reaction to any of the agents or any component used in this study.
10. Presence or suspicion of fungal, bacterial, viral, or other infection that is uncontrolled or requiring intravenous (IV) antimicrobials for management.
11. Uncontrolled or active infectious diseases, such as human immunodeficiency virus (HIV) infection, acute or chronic active hepatitis B or C, epstein-barr virus (EBV), and cytomegalovirus (CMV) infection.
12. History or presence of CNS disorder such as seizure disorder, cerebrovascular ischemia/hemorrhage, dementia, cerebellar disease, or any autoimmune disease with CNS involvement.
13. Subjects with cardiac atrial or cardiac ventricular lymphoma involvement.
14. History of myocardial infarction, cardiac angioplasty or stenting, unstable angina, or other clinically significant cardiac disease within 12 months of enrollment.
15. Expected or possible requirement for urgent therapy within 6 weeks due to ongoing or impending oncologic emergency (eg, tumor mass effect, tumor lysis syndrome).
16. Primary immunodeficiency.
17. History of autoimmune disease (e.g. Crohn's, rheumatoid arthritis, systemic lupus) resulting in end organ injury or requiring systemic immunosuppression/systemic disease modifying agents within the last 2 years.
18. History of symptomatic deep vein thrombosis or pulmonary embolism requiring systemic anticoagulation within 6 months of enrollment.
19. Any medical condition likely to interfere with assessment of safety or efficacy of study treatment.
20. Vaccine ≤ 6 weeks prior to planned start of conditioning regimen.
21. In the investigator's judgment, the subject is unlikely to complete all protocol-required study visits or procedures, including follow-up visits, or comply with the study requirements for participation.

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-02-15 (Actual); Primary Completion 2027-02-15 (Estimated); Study Completion 2028-02-15 (Estimated)

PRIMARY OUTCOMES:
Phase 1: Incidence of adverse events (AE) defined as DLT | First infusion date of CAR-T cells up to 28 days
  DLT is defined as any AE related to the investigational drug that occurs within 28 days after administration of the allogeneic Power3 (SPPL3) knock-out CD19 CAR-T and meets any one of the criteria listed in the DLT criteria. The severity of AE will be assessed according to NCI-CTCAE v5.0. cytokine release syndrome (CRS) and immune cell-associated neurotoxicity syndrome (ICANS) will be evaluated according to the standards released by ASTCT in 2019. GvHD according to criteria defined by the Mount Sinai Acute GVHD International Consortium.
  * Grade 3 aGVHD that does not resolve to Grade 1 or 2 within 7 days, with the exception of isolated skin involvement aGVHD;
  * Grade 3 CRS that does not resolve to grade 2 or lower within 2 weeks;
  * Grade 3 ICANS lasting for ≥ 7 days;
  * Any Grade ≥ 4 aGVHD or CRS or ICANS;
  * Any other Grade ≥ 4 and Grade 3 AE related to the allogeneic Power3 (SPPL3) knock-out CD19 CAR-T that lasts for ≥ 14 days, except hematology toxicity.
Phase 1: RP2D | 12 months
  The RP2D was determined through phase 1 study.
Phase 2: Objective response rate (ORR) | 24 months
  Objective response definition: a molecular response (MRD < 10^-4 post treatment) assessed by multiparameter flow cytometry and/or qPCR, or a morphologic complete response (CR), or a CR with incomplete blood count recovery (CRi). ORR is defined as the proportion of patients who have achieved objective response assessed by investigators.
Phase 2: Overall Survival (OS) | 24 months
  OS is defined as the time from CAR-T cells infusion to the date of death. Subjects who have not died by the analysis data cutoff date will be censored at the last contact date.
Phase 2: Progression Free Survival (PFS) | 24 months
  PFS is defined as the time from the CAR-T cells infusion date to the date of disease progression assessed by investigators, or death any cause. Participants not meeting the criteria for progression by the analysis data cutoff date were censored at the last evaluable disease assessment date.

SECONDARY OUTCOMES:
Phase 1 and phase 2: Level of CAR-positive T cells circulating in blood over time | 12 months
  Number and copy number of CAR-T cells were assessed by number in peripheral blood. Blood samples were collected before and one year after cell infusion (until CAR-T cells were not detected for two consecutive times) to detect the number and copy number of CAR-T cells, and to evaluate the pharmacokinetics of CAR-T.
Phase 1 and phase 2: Level of CD19+ cells in peripheral blood | Up to 28 days after infusion
  The level of CD19+ cells in peripheral blood will be detected by flow cytometry.
Phase 1 and phase 2: Level of interleukin 6 (IL-6) in peripheral blood | Up to 28 days after infusion
  The level of IL-6 in peripheral blood will be detected by enzyme-linked immuno sorbent assay.
Phase 1: 3-month ORR | 3 months
  The definition of ORR has already been mentioned above
Phase 1: OS | 24 months
  The definition of OS has already been mentioned above
Phase 1: PFS | 24 months
  The definition of PFS has already been mentioned above
Phase 2: Incidence of AE | 24 months
  AE is defined as any adverse medical event from the date of enrollment to 24 months after CAR-T cells infusion.

OTHER OUTCOMES:
Phase 1: Level of donor-specific antibody (DSA) in blood. | 12 months
  DSA refers to the specific antibody produced in the recipient's body targeting donor antigens after receiving CAR-T cell infusion from healthy donors.
Phase 1: Level of human anti-mouse antibodies (HAMA) | 12 months
  The levels of human against murine scFv antibodies in blood

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - Biotherapeutic Department of Chinese PLA General Hospital, Beijing, Beijing Municipality
  - Department of Hematology, Chinese PLA General Hospital, Beijing
  - Department of Hematology, Peking Union Medical College Hospital, Beijing
  - Department of Hematology, Tianjin First Central Hospital, Tianjin
  - Immune Cell Therapy Center, Blood Disease Hospital, Chinese Academy of Medical Sciences, Tianjin